CLINICAL TRIAL: NCT06858852
Title: A Multicenter, Randomized, Double-blind, Etomidate Parallel Controlled Phase III Clinical Trial Was Conducted to Evaluate the Efficacy and Safety of Methoxyethyl Etomidate Hydrochloride for Sedation/Anesthesia During Gastroscopy/Colonoscopy
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Methoxyethyl Etomidate Hydrochloride for Sedation/Anesthesia During Gastroscopy/Colonoscopy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-26-HCl-302
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Gastroscopy; Colonoscopy
MeSH Terms: interventions — ET-26 compound; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ET-26 0.8mg group (Experimental): Experimental
  Interventions: Drug: ET-26HCl 0.8mg/kg group
- Etomidate group (Active Comparator): Active Comparator
  Interventions: Drug: Etomidate Injectable Product 0.3mg/kg group

INTERVENTIONS:
Drug: ET-26HCl 0.8mg/kg group — The initial dose was 0.8 mg/kg administered as a single IV infusion over a period of 1 minute ±5 seconds. If needed, up to 50% of the starting dose was increased (30-seconds ± 5-seconds bolus)
  Arms: ET-26 0.8mg group
Drug: Etomidate Injectable Product 0.3mg/kg group — The initial dose was 0.3 mg/kg administered as a single IV infusion over a period of 1 minute ±5 seconds. If needed, up to 50% of the starting dose was increased (30-seconds ± 5-seconds bolus)
  Arms: Etomidate group

SUMMARY:
A total of 270 subjects undergoing gastroscopy/colonoscopy were randomly assigned to the methoxetomidate hydrochloride group and the etomidate group according to the ratio of 2:1 with etomidate as the control group.Neither the investigators nor the subjects were aware of the group assignments. Screening assessments for all subjects will be completed within D-14 to D-2 before the first dose. For all subjects who received the investigational drug, they were required to return to the research center on D2-5 to complete the corresponding examination before being discharged from the group. Compared with etomidate, the efficacy and safety of Methoxyethyl Etomidate Hydrochloride for sedation/anesthesia in gastroscopy/colonoscopy were further evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing routine gastroscopy/colonoscopy;
2. age ≥ 18 and ≤ 75 years old, regardless of gender;
3. American Society of Anesthesiologists (ASA) grade I-III;
4. Body mass index (BMI) 18-30 kg/m2 (including the cut-off value) and body weight ≤100 kg;
5. Serum cortisol concentrations were either normal or abnormal but not clinically significant as judged by the investigator
6. Vital signs during screening:

   respiratory rate ≥10 and ≤24 times/min; Pulse oxygen saturation (SpO2) ≥95% while breathing air; Systolic blood pressure (SBP) ≥90mmHg and ≤160mmHg; Diastolic blood pressure (DBP) ≥60mmHg and ≤100mmHg; Heart rate (ECG) ≥55 and ≤100 beats/min;
7. Able to understand the procedures and methods of this study, willing to sign the informed consent and strictly abide by the trial protocol to complete the study.

Exclusion Criteria:

1. patients with possible gastroduodenal outflow obstruction with retention of contents or upper gastrointestinal bleeding;
2. patients who were known or suspected to have allergies or contraindications to the components of the investigational drug or the prescribed regimen, or who were suspected to have epilepsy or severe liver and kidney dysfunction;
3. Predicted difficulty in intubation or ventilation (modified Markov score level III, level IV);
4. having any of the following respiratory management risks before/at the time of screening: 1) history of asthma, wheezing; 2) sleep apnea syndrome;
5. QTcF≥450 ms (male) or ≥470 ms (female) at screening and confirmed by review; Or clinically significant electrocardiographic abnormalities that were deemed by the investigator to be ineligible for the study;
6. use of any of the following drugs or treatments before screening:1) enrolled in a clinical trial of any drug within 1 month before screening; 2) use of medications or treatments that affect cortical function within 3 days before screening; 3) Use of medications that may affect QT interval within 2 weeks before screening;
7. During the screening period, the laboratory examination indicators exceeded the abnormal level and had clinical significance, and were not suitable for enrollment after evaluation by the investigators;
8. pregnant and lactating women; The reluctance of women or men of childbearing potential to use contraception for the entire dosing period; Subjects (including male subjects) who plan to become pregnant within 3 months after the trial;
9. Subjects with any other factors considered by the investigator to be ineligible for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of gastroscopy/colonoscopy | Within approximately 1 hour after injection
  From the time of bolus administration to the completion of gastroscopy/colonoscopy, the following two conditions were met simultaneously: (1) the number of additional doses within any 15 minutes was ≤5; (2) no use of rescue drugs.

SECONDARY OUTCOMES:
Sedation/anesthesia success rate | Within approximately 1 minute of the end of the injection
  Percentage of subjects with a MOAA/S score ≤1 after initial dosing of the investigational drug
Duration of successful sedation/anesthesia | within approximately 1minute after injection
  The time from the first administration of the experimental drug to the MOAA/S score ≤1
Duration from successful insertion to full consciousness | after approximately 30 minutes of the completion of the last injection
  the time from successful insertion to full awakening (the first time of three consecutive MOAA/S scores reaching 5 points
Duration from completion of experimental drug administration to full recovery | Within approximately 50 minutes of the completion of the last injection
  The time between the completion of the last trial drug administration and the subject's full recovery (the first of three consecutive MOAA/S scores of 5
The time from the end of treatment to full consciousness | Within approximately 60 minutes of the completion of the first injection
  The time from gastroscopy/colonoscopy withdrawal until the subject is fully awake (the first of three consecutive MOAA/S scores of 5
The time from the end of the endoscopic session to discharge from the room | A maximum of 10 minutes after awakening
  The first occurrence time from gastroscopy/colonoscopy withdrawal to 3 consecutive departures with Aldrete score ≥9
Rate of use of remedial drugs | 60minutes after injection
  Percentage of subjects who had used the sedative/anesthetic remedy propofol injection once or more
Test drug additions | 30minutes after injection
  the additional situation and dosage of drugs were summarized
Assessment of orientation | 20 minutes after the end of endoscopic treatment
  Orientation was evaluated when MOAA/S reached 5 points for the first time after the complete withdrawal of gastroscopy/colonoscopy
Anesthesiologists' satisfaction with the recovery state of the subjects was evaluated | 60 minutes after the end of endoscopic treatment
  The total score is 10, that is, a score of 0 indicates very dissatisfied and a score of 10 indicates very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Mengchang Yang, Principal Investigator — Sichuan Academy of Medical Sciences; Jin Liu, Principal Investigator — West China Hospital
Locations (6):
- China (6):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences · Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Guangyuan First People's Hospital, Guangyuan, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan